CLINICAL TRIAL: NCT05943223
Title: Assessing the Longitudinal Outcomes of Piperacillin/Tazobactam Versus ceftriAxone and Metronidazole for Children With Perforated Appendicitis (ALPACA): a Randomized Controlled Trial
Brief Title: Piperacillin/Tazobactam Versus ceftriAxone and Metronidazole for Children With Perforated Appendicitis (ALPACA)
Acronym: ALPACA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael Livingston, Pediatric Surgeon, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: McmasterCH
Record Dates: First submitted 2023-06-26; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Appendicitis Perforated
Keywords: Child; Piperacillin; Ceftriaxone; Metronidazole
MeSH Terms: conditions — Appendicitis | interventions — Piperacillin, Tazobactam Drug Combination; Saline Solution; Ceftriaxone; Metronidazole

STUDY DESIGN:
Intervention Model Description: Internal pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piperacillin/tazobactam (Experimental)
  Interventions: Drug: Piperacillin/tazobactam; Drug: Normal saline
- Ceftriaxone and metronidazole (Active Comparator)
  Interventions: Drug: CefTRIAXone Injection; Drug: Metronidazole Injection

INTERVENTIONS:
Drug: Piperacillin/tazobactam — Post-operative piperacillin/tazobactam 100 mg/kg IV q8h (to a maximum of 4.5 g IV q8h)
  Arms: Piperacillin/tazobactam
Drug: Normal saline — Post-operative normal saline 50 mL once daily
  Arms: Piperacillin/tazobactam
Drug: CefTRIAXone Injection — Post-operative ceftriaxone 50 mg/kg IV once daily (to a maximum of 2 g IV once daily)
  Arms: Ceftriaxone and metronidazole
Drug: Metronidazole Injection — Post-operative metronidazole 10 mg/kg IV q8h (to a maximum of 500 mg IV q8h)
  Arms: Ceftriaxone and metronidazole

SUMMARY:
This study is an internal pilot for a multicenter, blinded randomized controlled trial. The purpose of the multicenter trial is to determine whether post-operative piperacillin/tazobactam is more effective than ceftriaxone and metronidazole for children treated with laparoscopic appendectomy for perforated appendicitis. We plan to conduct an internal pilot study to determine whether a blinded multicenter randomized controlled trial is feasible.

DETAILED DESCRIPTION:
Acute appendicitis is the most common indication for emergency surgery in children. The management of this condition is typically an urgent laparoscopic appendectomy under general anesthesia. If the appendix is found to be perforated at the time of surgery, then patients need to stay in hospital for intravenous antibiotics. Patients who do not respond to antibiotic therapy experience prolonged length of stay, need for additional procedures (such as percutaneous drain insertion), or other complications. This represents significant morbidity for patients and their families.

Children with perforated appendicitis were previously treated with post-operative ampicillin, gentamicin, and metronidazole (also known as "triple therapy"). In 2008, a randomized controlled trial showed that triple therapy is non-inferior to ceftriaxone and metronidazole (CM) in terms of intra-abdominal abscess formation and wound infection. CM is also less expensive and has a simplified dosing regimen. As such, post-operative CM became the standard of care for perforated appendicitis at most children's hospitals.

In 2021, an open-label RCT suggested that piperacillin/tazobactam (PT) is more effective than CM for children with perforated appendicitis. Patients randomized to PT had a reduced rate of intra-abdominal abscess formation compared to those treated with CM (odds ratio (OR) 4.80, p=0.002). This trial was not blinded and there was no allocation concealment. In contrast, a multicenter, observational study reported no difference in the rate of intra-abdominal abscess formation among patients treated with PT compared to CM. The conflicting results of these two studies add further uncertainty regarding the choice of antibiotics for these patients.

Another factor that should be considered regarding the use of PT versus CM in children with perforated appendicitis is antibiotic stewardship. PT is a broad-spectrum antibiotic with increased effectiveness against Pseudomonas aeruginosa and resistant Escherichia coli. As a result, this medication is often reserved for patients with confirmed Pseudomonas infection, oncology patients with febrile neutropenia, or those who are critically ill and admitted to the intensive care unit.

The current study is an internal pilot for a multicenter, blinded randomized controlled trial. The purpose of the multicenter trial is to determine whether post-operative piperacillin/tazobactam is more effective than ceftriaxone and metronidazole for children treated with laparoscopic appendectomy for perforated appendicitis. We plan to conduct an internal pilot study to determine whether a blinded multicenter randomized controlled trial is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic appendectomy
* Perforated appendicitis confirmed intra-operatively (i.e., visible hole in appendix, fecalith found in peritoneal cavity, intra-abdominal abscess, and/or purulent fluid in peritoneal cavity)

Exclusion Criteria:

* Non-operative treatment (e.g., due to abscess)
* Interval laparoscopic appendectomy
* Conversion to open procedure
* Non-perforated appendicitis
* Confirmed or suspected allergy to penicillins or cephalosporins
* Renal impairment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Length of stay | Index admission
  Length of stay in hospital during index admission

SECONDARY OUTCOMES:
Percutaneous drain insertion | Within 30 days of surgery
  Percutaneous drain insertion by Interventional Radiology
Deep or organ-space surgical site infection | Within 30 days of surgery
  Deep or organ-space surgical site infection
Insertion of Peripherally Inserted Central Catheter (PICC) | Within 30 days of surgery
  Insertion of Peripherally Inserted Central Catheter (PICC)
Parenteral nutrition | Within 30 days of surgery
  Need for parenteral nutrition
Post-operative ultrasound | Within 30 days of surgery
  Need for post-operative ultrasound
Clostridium difficile infection | Within 30 days of surgery
  Clostridium difficile infection (confirmed with stool sample and requiring treatment)
Return to the emergency department | Within 30 days of surgery
  Return to the emergency department within 30 days of surgery
Readmission to hospital | Within 30 days of surgery
  Readmission to hospital within 30 days of surgery
Late complications | Telephone call 3 months after surgery
  Telephone confirmation of no additional complications related to perforated appendicitis requiring assessment in clinic, emergency department visit, or admission to hospital
Exit survey | Telephone call 3 months after surgery
  Parents will complete a descriptive questionnaire about the study by telephone

OTHER OUTCOMES:
Recruitment rate | Through study completion (average of 1 year)
  Number of participants randomized per month
Consent rate | Through study completion (average of 1 year)
  Number of participants who consent to participate divided by those who are approached for consent
Rate of protocol violations | Through study completion (average of 1 year)
  Number of participants who do not receive study treatments within 8 hours of surgery, miss a scheduled study treatment, and/or experience treatment crossover divided by those randomized
Rate of loss to follow-up | Through study completion (average of 1 year)
  Number of participants who cannot be contacted by phone 3 months after discharge from hospital divided by those randomized
Cost of trial | Through study completion (average of 1 year)
  Total cost of internal pilot study in Canadian dollars divided by the number of participants randomized

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Livingston, MD, MSc, Principal Investigator — McMaster Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St Peter SD, Snyder CL. Operative management of appendicitis. Semin Pediatr Surg. 2016 Aug;25(4):208-11. doi: 10.1053/j.sempedsurg.2016.05.003. Epub 2016 May 10. PMID 27521710
- [Background] Linnaus ME, Ostlie DJ. Complications in common general pediatric surgery procedures. Semin Pediatr Surg. 2016 Dec;25(6):404-411. doi: 10.1053/j.sempedsurg.2016.10.002. Epub 2016 Oct 29. PMID 27989365
- [Background] St Peter SD, Tsao K, Spilde TL, Holcomb GW 3rd, Sharp SW, Murphy JP, Snyder CL, Sharp RJ, Andrews WS, Ostlie DJ. Single daily dosing ceftriaxone and metronidazole vs standard triple antibiotic regimen for perforated appendicitis in children: a prospective randomized trial. J Pediatr Surg. 2008 Jun;43(6):981-5. doi: 10.1016/j.jpedsurg.2008.02.018. PMID 18558169
- [Background] Lee J, Garvey EM, Bundrant N, Hargis-Villanueva A, Kang P, Osuchukwu O, Dekonenko C, Svetanoff WJ, St Peter SD, Padilla B, Ostlie D. IMPPACT (Intravenous Monotherapy for Postoperative Perforated Appendicitis in Children Trial): Randomized Clinical Trial of Monotherapy Versus Multi-drug Antibiotic Therapy. Ann Surg. 2021 Sep 1;274(3):406-410. doi: 10.1097/SLA.0000000000005006. PMID 34132703
- [Background] Kashtan MA, Graham DA, Melvin P, Hills-Dunlap JL, Anandalwar SP, Rangel SJ. Ceftriaxone with Metronidazole versus Piperacillin/Tazobactam in the management of complicated appendicitis in children: Results from a multicenter pediatric NSQIP analysis. J Pediatr Surg. 2022 Oct;57(10):365-372. doi: 10.1016/j.jpedsurg.2021.11.009. Epub 2021 Nov 20. PMID 34876294
- [Background] Gerber JS, Jackson MA, Tamma PD, Zaoutis TE; COMMITTEE ON INFECTIOUS DISEASES, PEDIATRIC INFECTIOUS DISEASES SOCIETY. Antibiotic Stewardship in Pediatrics. Pediatrics. 2021 Jan;147(1):e2020040295. doi: 10.1542/peds.2020-040295. PMID 33372120
- [Derived] Briatico D, Safa N, Flageole H, Khan S, Pernica J, Eltorki M, Cohen E, Livingston MH. Assessing the Longitudinal outcomes of Piperacillin/tazobactam versus ceftriAxone and metronidazole for Children with perforated Appendicitis (ALPACA): A protocol for a pilot randomized controlled trial. PLoS One. 2025 Nov 7;20(11):e0335991. doi: 10.1371/journal.pone.0335991. eCollection 2025. PMID 41202087